CLINICAL TRIAL: NCT06846060
Title: The Effect of a Mindfulness-Based Self-Compassion Program Applied to Women Diagnosed With Breast Cancer on Spiritual Well-Being and Self-Compassion Levels: A Randomized-Controlled Study
Brief Title: A Mindfulness-Based Self-Compassion Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Haci Bektas Veli University (Other)
Responsible Party: Principal Investigator, Semra seyhan Şahin, RESEARCH ASSISTANT DR, Nevsehir Haci Bektas Veli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NEVU-NRS-SS-02
Record Dates: First submitted 2025-02-15; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Survivor
Keywords: breast cancer; minfulness; spiritual well-being; self-compassion
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): A mindfullness-based intervention program consisting of 8 sessions will be applied to the Intervention Group Awareness program intervention programs (Mindfullness) are a special comprehensive program that integrates the body and mind and consists of payments related to temporary local treatment of current yoga, diversity and awareness of the moment. According to the literature, the self-compassion program kept at home for 8-year-olds consists of 8 recordings in total, two recordings per week in groups of 8 people. He has goals and objectives specific to his personal record and yet there is a separate relationship day with the subject of his one information.
  Interventions: Behavioral: Mindfulness-Based Self-Compassion Program
- Control group (No Intervention): No intervention will be applied to the control group. Before and after the intervention program, the Coopersmith Self-Esteem Scale (GISS) and Spiritual Well-Being Scale (FACIT-SP-12) will be applied to the cotra group simultaneously with the experimental group.

INTERVENTIONS:
Behavioral: Mindfulness-Based Self-Compassion Program — Mindfulness-based intervention programs are a program that includes a special session in which body and mind are integrated, and consists of homework for participants on yoga, meditation and a mindfulness-based approach to vital events in order to be aware of the moment. The conscious awareness-based self-compassion program, created in line with the literature, consists of 8 sessions in total, in groups of 5-8 people, on the same day and time every week. There are specific goals and objectives for each session, and each session also has a separate theme along with its subject.
  Arms: intervention group

SUMMARY:
The purpose of this study is a pre-test-post-test, randomized controlled experimental study with a control group, planned to examine the effect of the mindfulness-based self-compassion program applied on women with breast cancer on spiritual well-being and self-compassion levels.

DETAILED DESCRIPTION:
The research was designed experimentally. The research will be conducted between February 2025 and April 2025 with female patients diagnosed with breast cancer who were treated in the oncology service of Cumhuriyet University Faculty of Medicine hospital in Sivas-Central province in the middle of Turkey and who meet the inclusion criteria. The study will be carried out face to face after obtaining the necessary institutional permissions. Participants to be included in the research will be included in the sample by taking into account the inclusion criteria at each stage. After the subject, purpose and method of the study are explained to the participants to be included in the study, they will be asked to fill out the informed consent form. Participants will then be divided into intervention and control groups by simple randomization method. Before the intervention, an information form, Self-Compassion Scale and Spiritual Well-Being Scale (FACIT-SP-12) will be applied to both groups. The implementation of the study will be carried out at the patient's convenience, in a time period that will not interfere with his treatment in any way, and in a special area determined by the hospital management, while preserving his privacy. A mindfullness-based intervention program consisting of 8 sessions will be applied to the Intervention Group. No intervention will be applied to the control group. At the end of the intervention program, the Self-Compassion Scale and Spiritual Well-Being Scale (FACIT-SP-12) will be administered to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast cancer,
* Women who are aware that they have been diagnosed with breast cancer,
* Women who volunteer to participate in the study,
* Women over the age of 18 with sufficient communication skills

Exclusion Criteria:

* Being diagnosed with any mental illness

Min Age: 18 Days | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women diagnosed with breast
Enrollment: 64 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-07 (Estimated)

PRIMARY OUTCOMES:
Coopersmith Self-Esteem Scale (CSES) | 5 week
  Turan and Tufan (1987) adapted the scale developed by Stanley Coopersmith (1967) into Turkish. Coopersmith (1967) found the reliability coefficient of the scale to be 0.91 for women and 0.80 for men. Additionally, the Cronbach Alpha coefficient of the scale was determined as 0.86. Each item of the scale, which consists of 25 items, is determined according to two options: "Suitable for me" and "Not suitable for me". The scoring of the scale is "4" for each correct statement and "0" for each incorrect statement; the highest score that can be obtained from the scale is 100 and the lowest score is 0. As the score obtained from the scale increases, individuals' self-esteem also increases. On the scale, a self-esteem level below 50 points is considered low, and a self-esteem level of 50 points and above is considered high. There are no reverse coded items in the scale.

SECONDARY OUTCOMES:
Spiritual Well-Being Scale (FACIT-SP-12) | 5 week
  The validity and reliability of the Spiritual Well-Being Scale (FACIT-Sp29 12), which was developed by Peterman et al. (2002) to measure the spiritual well-being of the individual in all chronic diseases, including cancer, was conducted in our country by Aktürk et al. (2017). The scale, which has 3 sub-dimensions (Meaning, Peace and Faith), allows the examination of all components of spiritual well-being. The scale is Likert type and consists of 12 items. The items in the scale have a numbering system from 0 to 4 (0-Not at all, 4-Extremely). The total score of the "Meaning" sub-dimension (Items 2,3,5,8) varies between 0 and 16 points, the total score of the "Peace" sub-dimension (Items 1,4,6,7) varies between 0 and 16 points, and the total score for the "Belief" sub-dimension (Items 9,10,11,12) varies between 0 and 16 points. The total scale score varies between 0 and 48. Higher scale values indicate greater spiritual well-being. In the study conducted by Aktürk (2017) on validity a

CONTACTS AND LOCATIONS:
Overall Officials: SEMRA SEYHAN SAHİN, Dr., Principal Investigator — Nevsehir Haci Bektas Veli University
Locations (1):
- Cumhuriyet University Medical Faculty Hospital, Sivas, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No